CLINICAL TRIAL: NCT04949451
Title: Time Restricted Feeding Intervention for Muscle and Metabolic Health (TRIMM)
Brief Title: Time Restricted Feeding, Muscle, and Metabolism
Acronym: TRIMM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TRIMM062021
Record Dates: First submitted 2021-06-16; First posted 2021-07-02 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TRF-C (Placebo Comparator): Follows time restricted feeding protocol.
  Interventions: Other: Control group - time restricted feeding only
- TRF-P (Experimental): Follows time restricted feeding protocol, consumes protein supplement
  Interventions: Dietary Supplement: Whey protein supplement
- TRF-S (Experimental): Follows time restricted feeding protocol, consumes ketogenic supplement
  Interventions: Dietary Supplement: Ketogenic aid

INTERVENTIONS:
Dietary Supplement: Whey protein supplement — Participants consume whey protein at the beginning of the eating period.
  Arms: TRF-P
Dietary Supplement: Ketogenic aid — Participants consume ketogenic aid upon waking.
  Arms: TRF-S
Other: Control group - time restricted feeding only — Time restricted feeding.
  Arms: TRF-C

SUMMARY:
Effective nutrition strategies for combatting and/or preventing obesity still need to be identified. This has been the case despite the numerous and different approaches that have been taken. Potential targets for combatting/preventing obesity have been identified, but long-term solutions have not emerged. This study uses time restricted feeding to study the role of dietary protein in obesity prevention and/or treatment. The objectives are to determine the role of skeletal muscle mass as a driver of energy-sensing mechanisms and peripheral signals that regulate appetite and energy intake in overweight and obese adults and to determine the effects of protein timing on muscle mass to regulate appetite and energy intake in overweight and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Resides in Northwest Arkansas
* Age 25-50 years
* BMI > 25
* All ethnicities
* Female and male

Exclusion Criteria:

* Food allergies
* Pregnant or breastfeeding
* Dietary restrictions (e.g. vegetarian, vegan, etc.)
* Trying to lose weight in last 3 months
* Pre-existing health conditions related to obesity (e.g. cardiovascular disease, diabetes, hypertension)
* Prescription medications related to heart disease or type 2 diabetes
* Fear of needles
* Smoker or vaping
* Currently taking protein supplements or other nutritional supplements which may interfere with study outcomes
* Consumes >4 alcoholic beverages per week

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-06-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Body composition | Change is being assessed at baseline and final day (day 120) of the intervention.
  Body composition measured using dual x-ray absorptiometry to determine the ration of lean/fat-free mass to fat mass.

SECONDARY OUTCOMES:
Whole body protein turnover | Change is being assessed at baseline and final day (day 120) of the intervention.
  Whole body protein turnover will be measured using 15N-alanine
Muscle mass | Change is being assessed at baseline and final day (day 120) of the intervention.
  Muscle mass will be measured using D3-creatine
Body weight | Change is being assessed at baseline, 4, 8, and 12 weeks.
  Body weight will be measured in kilograms.
Sleep | Change is being assessed at baseline and 12 weeks
  Sleep will be assessed using wrist Actigraphy for sleep duration and total time in bed.
Sleep Quality | Change is being assessed at baseline, 4, 8, and 12 weeks
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index survey
Mood | Change is being assessed at baseline, 4, 8, and 12 weeks
  Mood will be assessed using the Profile of Mood States Questionnaire
Grit | Change is being assessed at baseline, 4, 8, and 12 weeks
  Grit will be assessed using the grit questionnaire.
Self-reported physical activity | Change is being assessed at baseline, 4, 8, and 12 weeks
  Physical activity will be measured using the iPAQ survey
Dietary intake | Change is being assessed at baseline, 4, 8, and 12 weeks
  Dietary intake will be measured using weighed, 3-day food records
Fasting glucose | Change is being assessed at baseline, 4, 8, and 12 weeks
  Glucose will be measured as mg/dl
Hand grip | Change is being assessed at baseline, 4, 8, and 12 weeks
  Hand grip will be measured using a dynamometer.
Amino acids and metabolites | Change is being assessed at baseline, 4, 8, and 12 weeks
  Blood will be collected and plasma amino acids and metabolites will be assessed using commercially available kit for amino acid analysis for all circulating amino acids.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided